CLINICAL TRIAL: NCT00839137
Title: Exercise Therapy for Asthma (ETA Trial)
Acronym: ETA
Status: Terminated | Type: Observational
Why Stopped: Study proved difficult to recruit
Sponsor: Ohio State University (Other)
Responsible Party: Sponsor
Other Study IDs: 2003H0213
Record Dates: First submitted 2009-02-06; First posted 2009-02-09 (Estimated); Last update posted 2021-11-08 (Actual); Status verified 2021-11

CONDITIONS: Asthma
Keywords: asthma; exercise therapy
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- no exercise program group: group will continue with current level of activity and will be asked not to start an exercise program. They will be seen in the clinic three times a week for 12 weeks. These visits will be very brief; blood pressure, heart rate, oxygen level and peak flow will be measured at each visit
- exercise group: will meet three times a week for 12 weeks, following specific exercise program

SUMMARY:
The purpose of the study is to determine if a program of regular exercise can help reduce asthma symptoms and also reduce the inflammation caused by asthma. If successful, this would allow regular exercise to be recommended as a therapy for people with asthma, which could possibly reduce the amount of medicine that people with asthma need to control their asthma symptoms.

DETAILED DESCRIPTION:
This is a randomized, controlled, parallel-design study of the effectiveness of exercise therapy as add-on therapy in the treatment of mild to moderately severe asthma.

105 men and women between the ages of 18-50 years with asthma will be randomly assigned to one of two treatment groups: exercise therapy or control. The exercise therapy protocol is detailed below. The control group will receive usual asthma care. The control group will be instructed to maintain their current sedentary activity level, i.e. not to begin a formal or informal exercise program. In order to standardize contact with study personnel between the two groups the control group will be seen three times a week for clinic visits (exercise group will have sessions three times a week). The primary outcome measures are asthma control (asthma symptom score) and asthma-related inflammation. Secondary outcomes include exacerbation rate, asthma-related quality of life, generic quality of life, lung function, airways hyper-reactivity, and cardiovascular fitness. The effect of exercise therapy on inflammatory markers in blood, and sputum will be assessed by comparing results obtained at study completion versus those obtained at baseline.

ELIGIBILITY:
Inclusion Criteria:

* • 18-50 years old

  * 50 + years old with prior approval to begin an exercise program from primary care physician within 6 months of enrollment
  * Men and women

Asthma:

* Doctor diagnosed asthma
* Lung function tests must meet certain levels common in asthma patients
* Active, daily doctor-prescribed asthma controller medication (inhaled corticosteroid) for 2 months or longer at a minimum dose equivalent to fluticasone 88 mcg/day, about two (2) puffs. (you can be on other drugs as long as they are in the same dose range as fluticasone)
* Poor asthma control: Any one of the following conditions:

  * Use of beta-agonist (A bronchodilator medicine that opens the airways by relaxing the muscles around the airways that may tighten during an asthma attack )for asthma symptoms twice/week or more OR
  * Awakening from sleep with asthma symptoms more than once per week OR
  * One or more control problems identified on the Asthma Treatment and Control Questionnaire (ATAQ).

Smoking status:

* Non-smoker for 6 months or longer
* Less than 10 pack year (number of packs per day (x) years of smoking = pack years) smoking history

Exclusion Criteria:

* • Poor lung function

  * Current participation in a regular aerobic exercise program (formal or at home)
  * Any "yes" to any one of items a-e of question number two of the Stanford Usual Activity Questionnaire
  * Pregnancy
  * Sudden illness that accompanies fever (> 38.00 C or 100.40F) within 24 hours of Visit 2
  * Participation in another interventional research trial Other major chronic illnesses that would interfere with participation in the study

Medication use:

* Chronic oral corticosteroid use
* Oral corticosteroid use within 4 weeks of study start
* Anti-coagulants (An anticoagulant is a drug that helps prevent the clotting (coagulation) of blood.), insulin, any investigative drugs within 2 months

Drug allergy:

• Previous adverse effects from methacholine challenge

Non-adherence:

* Inability or unwillingness to provide consent
* Inability to perform aerobic exercise
* Inability to perform baseline measurements
* Less than 80% completion of screening period diaries
* Inability to contact by telephone
* Intention to move out of the area within 6 months

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: primary care clinic, community sample
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2003-12; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
To determine the effectiveness of a behavioral intervention, exercise therapy as a primary therapy for asthma | end of study
  To determine the effectiveness of a behavioral intervention, exercise therapy as a primary

SECONDARY OUTCOMES:
to determine how one program of exercise therapy affects asthma symptoms and inflammatory markers from the blood and the lung of asthmatics | end of study
  To determine the effectiveness of a behavioral intervention, exercise therapy as a primary

CONTACTS AND LOCATIONS:
Overall Officials: John G Mastronarde, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States